CLINICAL TRIAL: NCT06580665
Title: Randomized Clinical Trials Comparing Immunotherapy Plus Cryoablation (I-CA) Versus Cryoablation Alone for Stage I, Selected Stage IIa, Non-Small Cell Lung Cancer
Brief Title: Cryoablation with or Without Serplulimab in Treating Patients with Stage I-IIA Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Shanghai Henlius Biotech Co., Ltd. (Unknown); AccuTarget MediPharma (Shanghai) Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IS24040
Record Dates: First submitted 2024-08-11; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Cryoablation; Serplulimab; Early non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cryosurgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryoablation alone (CA group) (Experimental): Patients undergo cryoablation alone.
  Interventions: Procedure: Cryoablation
- Cryoablation combined with immunotherapy (I-CA group) (Experimental): Patients undergo cryoablation. If there are no significant postoperative complications, Serplulimab should be administered immediately. Cycles with Serplulimab repeat every 3 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Cryoablation; Drug: Serplulimab

INTERVENTIONS:
Procedure: Cryoablation — Patients undergo cryoablation.
Drug: Serplulimab — Patients undergo cryoablation. If there are no significant postoperative complications, Serplulimab should be administered immediately. Cycles with Serplulimab repeat every 3 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Arms: Cryoablation combined with immunotherapy (I-CA group)

SUMMARY:
Cryoablation is a minimally invasive technique that utilizes very low temperature to eliminate tumour cells for patients ineligible for surgery. It has been reported that cryoablation may enhance immune response and synergize with immunotherapy.

This study is a multicenter, randomized, controlled, exploratory trial, and is expected to enroll a total of 134 patients. The enrolled patients were stage Ia, Ib, or IIa lung cancer with negative driver gene mutations, who are considered high-risk for surgery or refuse surgery based on multidisciplinary evaluation. Eligible patients will be randomly assigned in a 1:1 ratio to receive either cryoablation alone (CA group) or cryoablation combined with immunotherapy (I-CA group). The study aims to evaluate the safety and clinical benefits of combining immunotherapy with cryoablation in the treatment of early-stage NSCLC by comparing progression-free survival (PFS), objective response rate (ORR), overall survival (OS), and the incidence of adverse events between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed as primary peripheral non-small cell lung cancer, preoperative staging suggested stage Ia, Ib, or IIa (size≤5 cm, T1-T2N0M0), according to the 9th edition of the TNM classification for lung cancer;
2. Negative driver gene mutation: driver genes were defined as EGFR, ALK, etc;
3. Age ≥18 years old;
4. The ECOG PS score is 0-2;
5. Expected survival ≥3 months;
6. Patients who are considered high-risk for surgery/radiotherapy or refuse surgery/radiotherapy based on multidisciplinary evaluation;
7. Patients who have not received previous immunotherapy with PD-1, PD-L1 or CTLA-4 antibodies;
8. All patients must agree to receive cryoablation (with or without Serplulimab) as an initial therapy and sign a study-specific consent form.

Exclusion Criteria:

1. Patients with poor cardiopulmonary function or other comorbidities who cannot tolerate multimode thermal therapy;
2. Patients whose chest CT indicated that the lung lesions could not be reached percutaneously or transbronchially;
3. Severe liver and kidney function and coagulation function abnormalities, platelet count <70×109/L;
4. Patients who have received other anti-tumor drugs in the past 6 months or have used immune checkpoint inhibitors before;
5. The patient has an uncontrolled disease (including but not limited to active infection, symptomatic congestive heart failure, unstable angina, arrhythmia, mental illness, etc.);
6. Primary immune deficiency or autoimmune diseases (e.g. rheumatoid arthritis, systemic lupus erythematosus, etc.);
7. Pregnant and lactating women;
8. Long-term use of steroid;
9. Other circumstances considered inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-08-11 (Estimated)

PRIMARY OUTCOMES:
3-year progression-free survival (PFS) | 3 years
  This refers to the length of time between the participant's first onset of disease progression or death from any cause after treatment.

SECONDARY OUTCOMES:
1-year, 2-year, and 3-year Objective Response Rate (ORR) | 3 years
  The percentage of patients that achieve complete response (CR) and partial response (PR) after treatment.
Overall Survival (OS) | 5 years
  The time from the start of treatment to the patient's death or the last follow-up, with a maximum observation period of 5 years from randomization.
Incidence of Adverse Events | 1 year
  Adverse events include those related to the cryoablation procedure occurring during or after the procedure, as well as drug-related adverse events caused by immunotherapy.
Potential Predictive and Immunological Biomarkers (lymphocyte phenotypes, PD-L1 expression, cytokines) | 1 year
  This refers to the changes from baseline in the immunological responses following the cryoablation (with or without Serplulimab) and comparison between the two groups, including the percentage and function of lymphocyte phenotypes, the expression of PD-L1, the concentration of IFN-γ levels, etc.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No